CLINICAL TRIAL: NCT06688357
Title: Revitalize Cognition: A Proof of Concept Study Using Transcranial Near Infrared Stimulation in Older Adults
Brief Title: Revitalize Cognition: Near Infrared Stimulation in Parkinson Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Parkinson's Disease Foundation (Other); The Parkinson's Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB201400128-A; 6AZ15 (Other Grant/Funding Number: FL DEPT OF HLTH ED ETHEL MOORE ALZHEIMER); PF-IMP-1938 (Other Grant/Funding Number: PARKINSONS FOU)
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
Keywords: Photobiomodulation; Near Infrared Light; Parkinson Disease; Neurostimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: randomized, sham controlled
Who Masked: Participant, Outcomes Assessor
Masking Description: The study is triple blinded. One of the co-investigators not involved in participant contact created a color-coded randomization schedule that mapped onto the active vs sham conditions. The randomization schedule was used to assign participants to one vs another color group. The devices were color coded. As such, the project coordinator, research assistants, and the PI were unaware of the participant's intervention status other than color assignment. All statistical analyses were done blindly using the color code for groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active NIR-PBM Parkinson Group (Active Comparator): The Active condition involves baseline testing, two weeks of Near Infrared-Photobiomodulation (NIR-PBM), and post-intervention testing. Cognitive, motor, mood, and neuroimaging outcomes are obtained before (baseline) and after the intervention. During outcome testing, Parkinson patients are evaluated "Off" their normal dopamine medications, following a standard 'overnight' washout. Otherwise, the PD patients were "ON" dopamine medications. The intervention consists of 6 sessions of NIR-photobiomodulation given 3 times/week for 2 weeks. During each session, NIR light is delivered via placement of six MedX LED superluminous diode clusters over the scalp for a total of 40 minutes. During stimulation, participants sit in front of a videomonitor and view nature documentaries (BBC Life series). This is done to standardize behavior during the intervention sessions.
  Interventions: Device: Active NIR-PBM (MedX 1116, MCT502)
- Sham NIR-PBM Parkinson Group (Sham Comparator): The Sham condition is identical in all respects to the Active condition except for use of a "sham" MedX device. The sham device was modified from the original MedX system to not deliver NIR light but was otherwise identical to the active device. Because NIR light is invisible, neither the participants nor interventionists can discern whether active or sham stimulation was being delivered. Otherwise, the Sham condition involved baseline testing (off medication), 2 weeks of sham NIR stimulation, and post-intervention procedures (Off dopamine medication).
  Interventions: Device: Sham NIR-PBM (MedX 1116, MCT502)

INTERVENTIONS:
Device: Active NIR-PBM (MedX 1116, MCT502) — Near infrared light was delivered using two MedX Rehab Console systems (MedX Health, 1116). Each MedX console included a control unit and 3 superluminous light emitting diode (LED) clusters. Each LED cluster (3MedX MCT502) consisted of 52 near infrared diodes and 9 visible red diodes. The 9 red diodes were deactivated. The energy delivered by each cluster was 1 joule [J]/cm2 in 45 sec at treatment wavelength of 870 nm per each 20 min. The LED cluster has an irradiance of 22.2 mW/cm2, treats an area of 22.48 cm2, with an energy density of 26.64/cm2 per cluster (total energy of 599J/cluster). During each session, the 6 clusters were arrayed on the scalp in 2 configurations, 20 minutes per array. Each configuration targeted 6 transcranial sites, guided by the 10-20 system, for a total of 12 sites during the 40-min session. Total energy delivered was 599J/cluster X 12 sites = 7188J. Dosing was based on a pilot study. This intervention was given 3 times/week for 2 weeks.
  Other Names: Transcranial Near Infrared Stimulation; Photobiomodulation
  Arms: Active NIR-PBM Parkinson Group
Device: Sham NIR-PBM (MedX 1116, MCT502) — The MedX sham intervention device is identical in all respects to the active device, except that the MedX console and diode clusters were modified to NOT deliver NIR light when turned on. The sham MedX devices were modified to deliver 'warmth', similar to that of the active devices. As with the active condition, a total of six sham interventions were given over a 2-week period, following the identical procedures described in the active condition.
  Other Names: Placebo
  Arms: Sham NIR-PBM Parkinson Group

SUMMARY:
The overall goal of this pilot, proof of concept study is to test a novel, relatively low cost, low risk and potentially high impact intervention for cognitive and motor symptoms associated with idiopathic Parkinson Disease. The intervention involves transcranial delivery of near infrared (NIR) light, aka as photobiomodulation (PBM). This pilot randomized controlled trial will examine whether NIR stimulation influences cognitive, mood, and motor symptoms in Parkinson patients relative to a sham treated group. The goal is to determine effect sizes for a potentially larger study.

Aims 1-3 of this study (Older Adult Specific) is registered separately under NCT02582593

DETAILED DESCRIPTION:
There are few validated approaches for minimizing cognitive changes that frequently accompany Parkinson disease (PD). The goal of this study is to test a novel and potentially high impact brain stimulation approach for enhancing cognitive, mood, and motor symptoms in individuals with PD. This brain stimulation approach involves transcranial delivery of near infrared (NIR) light, which is painless and undetectable, and enhances brain metabolism. This NIR stimulation approach is also known as photobiomodulation (PMB).

The study builds on the following premises:

Mitochondrial dysfunction has been implicated in both familial and nonfamilial Parkinson disease.

NIR stimulation is a novel intervention for enhancing mitochondrial energy metabolism; Indeed, research in cellular and animal models suggests that application of light in red (630-700nm) and near infrared wavelengths (808-904nm) is neuroprotective and improves mitochondrial function by promoting increased production of intracellular adenosine triphosphate (ATP), important for cellular metabolism and oxygenation.

Findings of positive effects of NIR stimulation on motor and cognitive symptoms in animal models of PD, both rodent and macaques. In these animal studies, strong evidence supports neuroprotective and 'rescue' effects of NIR stimulation from MPTP-induced neurodegeneration, including preservation of locomotor activity and midbrain dopaminergic neurons. It is unclear whether similar beneficial effects might be afforded humans with idiopathic Parkinson disease (PD).

As such, the goal is to conduct a proof-of-concept randomized control pilot study to determine feasibility, acceptability and efficacy of a NIR stimulation protocol in individuals with Parkinson disease (PD). The intervention will involve six sessions over a 2-week period, in which active or sham stimulation is applied to the head using a delivery system that has been approved as a nonsignificant risk since 2003. The delivery system involves six MedX superluminous light emitting diode clusters positioned on the head in distinct configurations for a total of 40 minutes of stimulation. Dosing was based on a pilot study. The investigators plan to enroll 24 non-demented individuals with PD who will be randomized to active or sham groups. Cognitive, motor, and mood outcomes will be obtained before and after the intervention. An exploratory aim involves neuroimaging changes (1P MRS, resting state fMRI). Outcomes will be obtained during the off-dopamine medication state (i.e., standard overnight withdrawal from dopamine medications). The investigators hope to learn whether NIR stimulation has potential for influencing motor and cognitive symptoms in individuals with PD, with goal of determining effect sizes for a potentially larger randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson disease by movement disorder neurologist using UK Brain Bank criteria
* Early-mid stage of disease severity
* Willingness to undergo baseline and post-intervention 'off' their normal dopamine medications
* Between 62 and 89 years of age
* Able to provide informed consent and perform cognitive and mood measures on a computer
* Willingness to be randomized to Sham or Real intervention
* Can devote 2 weeks to the intervention, and additional time for pre and post testing
* 8th grade education and ability to read on 8th grade level based on scores on the Wechsler Test of Adult Reading (WTAR) or the Wide Range Achievement Test-IV (WRAT-IV); ability to see 14 pt. text
* On stable doses of major medications for at least two months

Exclusion Criteria:

* History of brain abnormalities/ neurological disorders affecting cognition other than PD; No history of brain surgery
* Evidence of potential dementia based on cognitive screening (e.g., scores < 5th %ile on the Montreal Cognitive Assessement (MoCA) or the Dementia Rating Scale-2 (DRS-2) based on appropriate age, education and sex norms.
* Use of psychotics, sedatives or other medications with anticholinergic properties;
* Unstable or uncontrolled medical conditions (e.g.,HIV, severe kidney disease)
* Diagnosis of active cancer
* Use of photosensitive medications within 15 days of intervention
* Sensory loss (vision, hearing) or motor deficits that would preclude participation in the experimental cognitive tasks or neuropsychological assessment
* Current or past history of major psychiatric disturbance including schizophrenia, or active psychosis, bipolar disorder, current major depressive episode, current alcohol or substance abuse or history thereof within the past six months. The investigators are not excluding individuals who are taking antidepressants or anti-anxiety medications, however, use of antidepressants and anxiolytics will be recorded and data will be analyzed in post-hoc analyses
* Previous participation in a cognitive training study within the last six months

Ages: 62 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Bowers, PhD, Principal Investigator — The University of Florida
Locations (1):
- Norman Fixel Institute for Neurological Diseases, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified cognitive, mood, and motor data will be made available to other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available starting June 2026.
Access Criteria: Requesters must have IRB approval.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All Parkinson participants were recruited from the Fixel Institute of Neurological Disease at the University of Florida. Participants were recruited directly from clinics and/or from the INFORM database, an IRB approved database which includes individuals who agreed to be contacted by researchers for potential participation in ongoing IRB approved studies.
Pre-assignment Details: Of the 23 consented participants, seven were excluded and not randomized. This included two individuals who declined to participate due to requirement that they undergo pre and post intervention testing when they were 'off' their normal dopamine medications. Another five were excluded due to low scores on a cognitive screener (MoCA), high scores on a mood measure, and confounding medical comorbidities (i.e., TBI, stroke).
Groups:
- Active NIR-PBM Parkinson: In the ACTIVE NIR-PBM arm, Parkinson participants received 6 sessions of transcranial NIR-PBM over a 2-week period. Each session involved 40 minutes of active stimulation across a total 12 intracranial sites. Stimulation was delivered via use of a MedX console system involving six superluminous LED clusters positioned over the head.
- Sham NIR-PBM Parkinson: In the SHAM NIR-PBM arm, Parkinson participants underwent identical intervention procedures as those in the 'active' group. However, the sham MedX device did not deliver near infrared light when turned on. The Sham condition involved 6 sessions over a two-week period; each session involved 40 minutes of sham NIR stimulation using a modified MedX delivery system.
Period: Overall Study
Arm/Group | Active NIR-PBM Parkinson | Sham NIR-PBM Parkinson
Started | 8 | 8 (1 participant withdrew at the beginning of baseline testing due to inability to tolerate being "off" the normal dopamine medication. This person completed half of one cognitive measure, before stopping, and did not undergo any intervention.)
Completed | 8 | 7
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Parkinson Group - Active NIR-PBM: Parkinson participants randomized to the Active group underwent baseline testing, followed by 6 sessions of transcranial NIR-PBM over a 2-week period, and immediate followup testing. Outcome measures were obtained at baseline and followup. Each intervention session involved 40 minutes of active NIR stimulation across a total 12 intracranial sites. Stimulation was delivered via use of a MedX console system involving six superluminous LED clusters. The power density used was 500 milliwatts (mW) with a cumulative fluence (energy density) of 312 Joules/cm2 (26 J/cm2 applied at 12 sites).
- Parkinson Group - Sham NIR-PBM: Parkinson participants randomized to the Sham group underwent identical procedures as those in the 'active' group. However, during the intervention phase, the near infrared deliver device (MedX console) was modified and did not deliver NIR light when turned on. The Sham condition involved 6 intervention sessions over a 2-week period. Each session consisted of 40 minutes of sham NIR stimulation using a modified MedX delivery system.
- Total: Total of all reporting groups
Arm/Group | Parkinson Group - Active NIR-PBM | Parkinson Group - Sham NIR-PBM | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (5.53) | 68.8 (2.67) | 71.07 (4.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
MoCA [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) is a widely used cognitive screener for dementia that was administered prior to beginning the trial. The MoCA scale ranges from 0 to 30 points, with higher scores reflecting better cognition. Participant scores were screened using age, education, sex, and race based norms from >8300 older adults (Sachs et al., 2020).
  units on a scale | 25.2 (4.17) | 27.4 (3.2) | 26.4 (3.75)
Duration of Parkinson symptoms [Mean (Standard Deviation); unit: years] — This refers to duration of Parkinson motor symptoms in years.
  years | 7.75 (6.39) | 5.29 (2.21) | 6.6 (4.91)
Parkinson Subtype- Tremor Predominant [Count of Participants; unit: Participants] — This refers to number of Parkinson participants whose initial motor symptoms were characterized as primarily involving tremors (versus a non-tremor presentation involving motor rigidity). This is important as some research suggests that tremor predominant PD is associated with less rapid progression of cognitive and other symptoms.
  Participants
    Tremor Predominant | 6 | 5 | 11
    Akinetic Rigid | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Fluency Composite From NIH Examiner (Kramer et al., 2014).
Description: The Fluency Composite is derived from the NIH Examiner, a computer-based battery of executive functioning tasks (Kramer et al., 2014). This composite was chosen due to known verbal fluency difficulties in individuals with Parkinson Disease. Verbal fluency tasks in the NIH Examiner include 2 trials of letter fluency and 2 trials of semantic fluency which are combined to yield a Fluency Composite that ranges from -3.0 to 3.0; higher scores correspond to better fluency performance. A change score is calculated by subtracting the baseline scores from the post-test scores. Greater positive change scores mean better outcome.
Time Frame: Baseline and Post-Intervention (2 weeks)
Population: Participants included nondemented individuals with Parkinson disease who were randomized to active or sham intervention groups. During outcome testing, PD participants were "off" their normal dose of dopamine medication, following the standard overnight washout period.
Measure: Mean (Standard Deviation); unit: z-score
Groups:
- Parkinson Group - Active NIR-PBM: In this arm, Parkinson participants received 6 sessions of transcranial NIR-PBM over a 2-week period. Each session involved 40 minutes of active NIR stimulation across a total 12 intracranial sites. Stimulation was delivered via use of a MedX console system involving six superluminous LED clusters. The power density used was 500 milliwatts (mW) with a cumulative fluence (energy density) of 312 Joules/cm2 (26 J/cm2 applied at 12 sites).
- Parkinson Group - Sham NIR-PBM: In the SHAM arm, Parkinson participants underwent identical intervention procedures as those in the 'active' group. However, the sham MedX device did not deliver NIR light when turned on. The Sham condition involved 6 sessions over a two-week period. Each session involved 40 minutes of sham NIR stimulation using modified MedX delivery system that delivered no NIR light.
Arm/Group | Parkinson Group - Active NIR-PBM | Parkinson Group - Sham NIR-PBM
Number analyzed (Participants) | 8 | 7
z-score | 0.334 (0.374) | -0.0287 (0.354)
Statistical Analysis 1: Comparison: Parkinson Group - Active NIR-PBM vs Parkinson Group - Sham NIR-PBM; Independent sample t-test conducted to examine difference in pre-post intervention change scores for the active vs sham intervention groups. Cohen's d was calculated to determine effect size; Test type: Superiority; p = .077, t-test, 2 sided — t (13) = 1.920. Only 1 comparison with 2 means, thus no adjustment necessary; Cohen's d = 0.99

2. Primary Outcome: ARENA Spatial Navigation Memory Task-Learning Composite
Description: ARENA is a task of spatial memory-navigation that has been linked to hippocampal function and is a human analogue to the Morris water maze, which has shown sensitivity to NIR stimulation in Alzheimer's transgenic mice. ARENA requires participants to learn and navigate to a hidden target location in a simulated environment. It involves use of a joystick over a series of 8 learning trials and one final probe trial. On each learning trial, the path length and time to reach the target are recorded. The Learning dependent variable is a composite score consisting of mean z-scores for path length and for time to reach the target (Learning Composite). A change score is computed by subtracting the baseline Learning Composite from the post-intervention Learning Composite z-score. Higher scores mean a better outcome.
Time Frame: Baseline and Post-Intervention (2 weeks)
Population: Participants included nondemented individuals with Parkinson disease who were randomized to active or sham intervention groups. During outcome testing, PD participants were evaluated "off" their normal dose of dopamine medication, following the standard overnight washout period.
Measure: Mean (Standard Deviation); unit: z-score
Groups:
- Parkinson Group - Active NIR-PBM: In the ACTIVE arm, Parkinson participants received 6 sessions of active transcranial NIR-PBM over a 2-week period. Each session involved 40 minutes of active NIR stimulation across a total 12 intracranial sites. Stimulation was delivered via use of a MedX console system involving six superluminous LED clusters. The power density used was 500 milliwatts (mW) with a cumulative fluence (energy density) of 312 Joules/cm2 (26 J/cm2 applied at 12 sites).
- Parkinson Group - Sham NIR-PBM: In the SHAM arm, Parkinson participants underwent identical intervention procedures as those in the 'active' group. However, the sham MedX device did not deliver NIR light when turned on. The Sham condition involved 6 sessions over a 2-week period. Each session involved 40 minutes of sham NIR stimulation using a modified MedX delivery system.
Arm/Group | Parkinson Group - Active NIR-PBM | Parkinson Group - Sham NIR-PBM
Number analyzed (Participants) | 8 | 7
z-score | -0.1088 (1.06) | -0.8495 (0.799)
Statistical Analysis 1: Comparison: Parkinson Group - Active NIR-PBM vs Parkinson Group - Sham NIR-PBM; independent sample t-test; Cohen's d effect size; Test type: Superiority; p = .159, t-test, 2 sided — t(13) = 1.504; only 1 comparison of 2 values, thus no adjustment is necessary; Cohen's D = 0.779

3. Primary Outcome: ARENA Spatial Navigation Memory Task - Total Composite
Description: ARENA is a computer-based task of spatial memory-navigation that has been linked to hippocampal function and is a human analogue to the Morris water maze. ARENA consists of 9 learning trials and one final probe trial. On each learning trial, the path length and time to reach the target are recorded. On each probe trial, the percent time spent in the spatial quadrant where the target is located is recorded. The dependent variable is a total composite score consisting of mean z-scores for path length, time to reach the target, and %time in the target quadrant during the probe trial (Total Composite). A change score is computed by subtracting the baseline Total Composite z-score from the post-intervention Composite z scores. Higher scores mean better outcome.
Time Frame: Baseline and Post-Intervention (2 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Parkinson Group- Active NIR-PBM: In the ACTIVE arm, Parkinson participants received 6 sessions of transcranial NIR-PBM over a 2-week period. Each session involved 40 minutes of active NIR stimulation across a total 12 intracranial sites. Stimulation was delivered via use of a MedX console system involving six superluminous LED clusters. The power density used was 500 milliwatts (mW) with a cumulative fluence (energy density) of 312 Joules/cm2 (26 J/cm2 applied at 12 sites).
Arm/Group | Parkinson Group- Active NIR-PBM | Parkinson Group - Sham NIR-PBM
Number analyzed (Participants) | 8 | 7
units on a scale | -0.1750 (.91776) | -0.4478 (.5372)
Statistical Analysis 1: Comparison: Parkinson Group- Active NIR-PBM vs Parkinson Group - Sham NIR-PBM; independent samples t-test, cohen's d effect size; Test type: Superiority; p = .503, t-test, 2 sided — t (13) = 0.688; only 1 comparison, adjustment not necessary; df = 13; Cohen's D = 0.356

4. Primary Outcome: Gait Stride Length Variability
Description: Gait is assessed using the Primary Gait Screen (Schmidt et al., 2019) that requires participants to walk the length of an 8-meter pressure sensitive mat (Zeno Walkway, 120Hz, Zeno Metrics), turn around, and return to the beginning of the walkway. Gait variability during forward walking was selected because in PD, greater variability is associated with increased number of falls and is one of the most disabling symptoms in PD. For this outcome, variability in stride length is indexed by the individual's standard deviation (SD) of stride length measured in centimeters; higher SD scores indicate worse performance. A change score is calculated by subtracting baseline SD of stride length from the post-intervention scores. Negative change scores mean better performance, whereas positive change scores mean worse performance.
Time Frame: Baseline and Post-Intervention (2 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: standard deviation
Groups:
- Parkinson Group - Active NIR-PBM: In the ACTIVE arm, Parkinson participants received 6 sessions of transcranial NIR-PBM over a 2-week period. Each session involved 40 minutes of active NIR stimulation across a total 12 intracranial sites. Stimulation was delivered via use of a MedX console system involving six superluminous LED clusters. The power density used was 500 milliwatts (mW) with a cumulative fluence (energy density) of 312 Joules/cm2 (26 J/cm2 applied at 12 sites).
Arm/Group | Parkinson Group - Active NIR-PBM | Parkinson Group - Sham NIR-PBM
Number analyzed (Participants) | 8 | 7
standard deviation | -0.388 (1.097) | .854 (1.442)
Statistical Analysis 1: Comparison: Parkinson Group - Active NIR-PBM vs Parkinson Group - Sham NIR-PBM; Independent sample t-test used to examine pre-post intervention change scores in active vs sham groups; Cohen's d was calculated to estimate effect size; Test type: Superiority; p = 0.08, t-test, 2 sided — t(13) = 1.893; only one comparison of 2 scores, thus no adjustment for multiple comparisons was necessary; df = 13; Cohen's D = -.922

5. Secondary Outcome: Working Memory Composite From the NIH Examiner (Kramer et al., 2014)
Description: This Working Memory composite is derived from a computer-based battery of executive functioning tasks (NIH Examiner). This composite was chosen due to known working memory difficulties in individuals with Parkinson disease. The Working Memory composite consists of scores from the N-back task and a Dot Counting task, which are combined to yield a composite score that ranges from -3 to 3.0; higher scores correspond to better working memory. A change score is calculated by subtracting the baseline Working Memory Composite from the post-intervention Working Memory Composite.
Time Frame: Baseline and Post (2 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Parkinson Group - Active NIR-PBM | Parkinson Group - Sham NIR-PBM
Number analyzed (Participants) | 8 | 7
z-score | 0.1491 (0.1516) | -0.1253 (.4822)
Statistical Analysis 1: Comparison: Parkinson Group - Active NIR-PBM vs Parkinson Group - Sham NIR-PBM; independent sample t-test, Cohen d effect size; Test type: Superiority; p = .149, t-test, 2 sided — t (13) = 1.533; only 1 comparison, no adjustment necessary; Cohen's D = 0.793

6. Secondary Outcome: Rey Auditory Verbal Learning Test (RAVLT)
Description: The RAVLT is a commonly used memory task in clinical settings. It is a 15-item word list learning task given over 5 trials followed by delayed recall of the list 20-30 minutes later. The major outcome is number of items freely recalled after the delay. Scores can range from 0 to 16 (maximum number of words), with higher score reflecting better performance. A change score is calculated by subtracting the baseline score from the post-intervention score. Higher difference scores indicate better performance due to intervention.
Time Frame: Baseline and Post (2 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parkinson Group - Active NIR-PBM | Parkinson Group - Sham NIR-PBM
Number analyzed (Participants) | 8 | 7
score on a scale | 2.38 (2.446) | 0.57 (1.272)
Statistical Analysis 1: Comparison: Parkinson Group - Active NIR-PBM vs Parkinson Group - Sham NIR-PBM; independent sample t-test was used to examine difference in Post-Pre intervention change in the Active vs the Sham groups; Effect size was estimated using Cohen's d; Test type: Superiority; p = .104, t-test, 2 sided — t(13) = 1.749; only 1 comparison with 2 values, thus no adjustment for multiple comparisons; df = 13; Cohen's D = 0.905

7. Secondary Outcome: Negative Affect Scale From the Emotion Module of the NIH Toolbox
Description: The Negative Affect scale is derived from the emotion module of the NIH Toolbox, a 12-22 minute self-report assessment that surveys current emotion health. The Negative Affect Scale is based on ratings of a series of emotion words. Questions comprise Likert-type items using computerized adaptive testing based on item response theory, resulting in a normed T score (mean of 50, SD of 10). The Negative Affect scale includes items pertaining to fear, anger, sadness. Scores below 40T indicate low levels of negative affect and scores above 60T indicate higher levels of negative affect. A difference score is computed by subtracting the baseline score from the post-intervention score.
Time Frame: Baseline and Post-Intervention (2 weeks)
Population: Individuals with idiopathic Parkinson disease who were tested 'off' dopaminergic medications
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Parkinson Group - Active NIR-PBM: Parkinson participants assigned to the ACTIVE arm received 6 sessions of transcranial NIR-PBM over a 2-week period. Each session involved 40 minutes of active NIR stimulation across a total 12 intracranial sites. Stimulation was delivered via use of a MedX console system involving six superluminous LED clusters. The power density used was 500 milliwatts (mW) with a cumulative fluence (energy density) of 312 Joules/cm2 (26 J/cm2 applied at 12 sites).
Arm/Group | Parkinson Group - Active NIR-PBM | Parkinson Group - Sham NIR-PBM
Number analyzed (Participants) | 8 | 7
T-score | -1.95 (3.59) | -.922 (4.16)
Statistical Analysis 1: Comparison: Parkinson Group - Active NIR-PBM vs Parkinson Group - Sham NIR-PBM; independent sample t-tests examining Post-Baseline differences for the Active vs the Sham groups; Effect size computed using Cohen's d score; Test type: Superiority; p = .614, t-test, 2 sided — t(13) = -.516; only 1 comparison of 2 means, no adjustment needed; Cohen's D = -0.267

8. Other Pre Specified Outcome: Unified Parkinson Disease Rating Scale Motor Scale (Part III) - Off Dopamine Medication
Description: Part III of the Unified Parkinson Disease Rating Scale (UPDRS) is a standard clinical rating scale for motor symptoms in individuals with Parkinson disease. It is clinician administered by a trained rater and involves ratings of motor tremors, rigidity, and slowness. In the research setting, the scale is videotaped for later scoring by a trained rater who is blinded to group assignment. The Part III motor scale score ranges from 0 to 108 and involves 27 responses to 14 questions. Higher scores are worse and reflect more severe motor symptoms. A change score is computed by subtracting baseline UPDRS motor score from the post-intervention score. Greater change in negative direction reflects better outcome.
Time Frame: Baseline and Post-Intervention
Population: Patients with Parkinson disease who were tested "off" dopamine medication following standard overnight washout.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parkinson Group - Active NIR-PBM | Parkinson Group - Sham NIR-PBM
Number analyzed (Participants) | 8 | 7
score on a scale | -3.87 (5.22) | 0.43 (7.91)
Statistical Analysis 1: Comparison: Parkinson Group - Active NIR-PBM; independent samples t-test, effect size computation (cohen's d); Test type: Superiority; p = .230, t-test, 2 sided — t(13) = -1.260; only 1 comparison of 2 values, no need for adjustment; Cohen's D = 0.652

ADVERSE EVENTS:
Time Frame: 3 Weeks
Description: Does not differ
Groups:
- Parkinson Group NIR: Transcranial Near Infrared Stimulation for Parkinson's Disease participants who will attend a total of 6 treatment sessions over a two-week period. During each session, stimulation via light emitting diode clusters will occur for a total of 60 minutes. Four light emitting diode (LED) clusters will be applied in 3 distinct configurations. There will be 20 minutes of stimulation at each of these 3 configurations. Each configuration will target 4 sites, for a total of 12 sites over the course of the 60-minute session. The power density used will be 500 milliwatts (mW) with a cumulative fluence (energy density) of 312 Joules/cm2 (26 J/cm2 applied at 12 sites). It is estimated that approximately 6 Joules/cm2 will reach the cortex with each daily treatment.
  MedX 1116 Rehab Console: This intervention makes use of transcranially applied near infrared light using light emitting diodes. Near infrared light will be applied to the scalp for a period of 1 hour at each session. A total of six session will be held.
- Parkinson Group - Sham: Parkinson's Disease participants in the sham control group will undergo identical procedures as the intervention group - screening, baseline testing, and LED cluster placement procedures. However, during the near infrared (NIR) session, the MedX console will not be turned on and no active stimulation will be applied.
  Sham MedX 1116 Rehab Console: This intervention makes use of sham transcranially applied near infrared light using light emitting diodes. Light emitting diodes (but not near-infrared light) will be applied to the scalp for a period of 1 hour at each session. A total of six session will be held.
Arm/Group | Parkinson Group NIR | Parkinson Group - Sham
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parkinson Group NIR (N=8) | Parkinson Group - Sham (N=8)
Medication (Nervous system disorders) | 0 (0) | 1 (1) — Participant became agitated at the start of the baseline session & indicated they felt ill being off their normal dopamine medication. They asked to withdraw from the study. They had been randomized but had not started the intervention.

LIMITATIONS AND CAVEATS:
This trial was designed to assess feasibility and determine effect sizes for larger trial. Moving forward, the ARENA task is not an ideal memory measure in the PD cohort due to reliance on motor skills (i.e., using a joystick); this caveat is further amplified given that outcome testing took place when PD participants were "off" dopamine medications and thus experiencing more severe motor symptoms. This trial took place during COVID epidemic and resulted in smaller than hoped for sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT06688357/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-13): https://cdn.clinicaltrials.gov/large-docs/57/NCT06688357/SAP_001.pdf